CLINICAL TRIAL: NCT01925950
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of the Safety and Efficacy of orBec® (Oral Beclomethasone 17,21-Dipropionate) Administered as Monotherapy in the Treatment of Upper Gastrointestinal (GI) Symptoms Caused by GVHD in Patients With Chronic GI GVHD
Brief Title: Study of orBec® as Monotherapy in the Treatment of Patients With Upper GI Symptoms Caused by Chronic Graft Versus Host Disease (GVHD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to patient enrollment challenges.
Sponsor: Soligenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BDP-GVHD-08
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Results first posted 2018-10-04 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Chronic Gastrointestinal Graft vs Host Disease
Keywords: BDP; orBec; GVHD; beclomethasone dipropionate; bone marrow transplant; hematopoietic cell transplant; HCT; stem cell transplant; marrow transplant; SCT; beclomethasone 17,21-dipropionate
MeSH Terms: interventions — alpha-ketoisovalerate dehydrogenase phosphatase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Control
  Interventions: Drug: Placebo
- orBec (Experimental): Investigational drug
  Interventions: Drug: orBec

INTERVENTIONS:
Drug: orBec
  Other Names: oral BDP; oral beclomethasone 17,21-dipropionate
  Arms: orBec
Drug: Placebo
  Arms: Placebo

SUMMARY:
Use of an oral topically-active glucocorticoid with limited side effects may control the gastrointestinal inflammatory process of GVHD and minimize glucocorticoid exposure.

ELIGIBILITY:
Inclusion Criteria:

* Receipt of allogeneic hematopoietic cell transplant >100 days prior to consent
* Documented cGVHD as defined by the NIH consensus criteria in at least one organ system other than the GI tract (for example, cGVHD of the oral cavity would qualify as a criterion)
* Endoscopic findings consistent with GI GVHD
* Must be able to swallow tablets
* Must be able to read and understand informed consent
* Adequate birth control methods for the duration of the study

Exclusion Criteria:

* >500 mL/day of diarrhea on any 1 day within 3 days prior to the first dose of study drug
* GI infection
* Multi-organ failure or other condition that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* HIV seropositivity
* Pregnant or nursing female
* Use of any investigational drug to treat chronic GVHD within 28 days of the first dose of study drug
* Evidence of recurrent or progressing malignant disorder that was the indication for HCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo was formulated as 1 mg immediate release (IR) and 1 mg delayed release (DR) tablets, which comprised 1 dose of study drug.
  Part 1: 2 mg of placebo 4 times per day for up to 16 weeks.
  Part 2: Patients who achieved a Complete Response (CR) on Part 1 were to taper study drug according to the following schedule:
  Weeks 17-24: 2 mg placebo 3 times per day, up to 8 weeks; Weeks 25-32: 2 mg placebo 2 times per day, up to 8 weeks; Weeks 33-48: 2 mg placebo daily, up to 16 weeks.
- orBec: orBec, oral beclomethasone dipropionate, was formulated as 1 mg immediate release (IR) and 1 mg delayed release (DR) tablets, which comprised 1 dose of study drug.
  Part 1: 2 mg of orBec 4 times per day for up to 16 weeks.
  Part 2: Patients who achieved a Complete Response (CR) on Part 1 were to taper study drug according to the following schedule:
  Weeks 17-24: 2 mg orBec 3 times per day, up to 8 weeks; Weeks 25-32: 2 mg orBec 2 times per day, up to 8 weeks; Weeks 33-48: 2 mg orBec daily, up to 16 weeks.
Period: Part 1
Arm/Group | Placebo | orBec
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0
Period: Part 2
Arm/Group | Placebo | orBec
Started | 1 | 0 (The 1 orBec subject completed Part 1 but did not meet the criteria of a CR to continue to Part 2)
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Control
  Placebo
- orBec: Investigational drug
  orBec
- Total: Total of all reporting groups
Arm/Group | Placebo | orBec | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Gastrointestinal (GI) Graft-vs-Host Disease (GVHD) Symptoms
Description: Patients who achieved a Complete Response (CR) of their GI GVHD Symptoms during the Part 1, 16 week treatment period and who remained a CR at the end of the 16 week treatment period were to be eligible to continue into Part 2 of the study. All others were to discontinue.
  GI GVHD was assessed using a composite score based on the symptoms of satiety, nausea/vomiting, and anorexia. Each symptom was scored on a scale of 0-3, such that the minimum score = 0 and the maximum score = 9. At entry, all subjects must have a score of ≥ 3. A CR will be defined as a composite score of 0.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Matching placebo was formulated as 1 mg immediate release (IR) and 1 mg delayed release (DR) tablets, which comprised 1 dose of study drug.
  2 mg of placebo 4 times per day for up to 16 weeks.
- orBec: orBec, oral beclomethasone dipropionate, was formulated as 1 mg immediate release (IR) and 1 mg delayed release (DR) tablets, which comprised 1 dose of study drug.
  2 mg of orBec 4 times per day for up to 16 weeks.
Arm/Group | Placebo | orBec
Number analyzed (Participants) | 1 | 1
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 48-week study period
Arm/Group | Placebo | orBec
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=1) | orBec (N=1)
biliary strictures (Hepatobiliary disorders) | 1 (1) | 0 (0)
fungal pneumonia (Infections and infestations) | 1 (1) | 0 (0)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pulmonary emboli (Vascular disorders) | 1 (1) | 0 (0)
intractable pain (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days